CLINICAL TRIAL: NCT06864585
Title: Zavicefta Combination for Intravenous Infusion Special Investigation - Surveillance on Patients With Sepsis or Renal Impairment (Creatinine Clearance ≤ 50 mL/Min) -
Brief Title: A Study to Learn About the Study Medicine - Zavicefta in Patients With Sepsis or Loss of Kidney Function in Japan
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3591038
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Infectious Diseases
Keywords: Sepsis; Renal impairment; Zavicefta; Avibactam; Ceftazidime
MeSH Terms: conditions — Communicable Diseases; Sepsis; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Avibactam sodium/Ceftazidime hydrate: Patients with sepsis or renal impairment (creatinine clearance ≤ 50 mL/min) who are administrated with Zavicefta (Avibactam sodium/Ceftazidime hydrate) for the first time
  Interventions: Drug: Avibactam sodium/Ceftazidime hydrate

INTERVENTIONS:
Drug: Avibactam sodium/Ceftazidime hydrate — The recommended adult dosage is 2.5 g (0.5 g of avibactam and 2 g of ceftazidime) administered by intravenous infusion over a period of 2 hours 3 times daily. For peritonitis, intra-abdominal abscess, cholecystitis, and liver abscess, Zavicefta should be co-administered with a metronidazole injection.
  Other Names: Zavicefta

SUMMARY:
The purpose of this study is to learn about the safety and how effective is Zavicefta under actual clinical practice in Japan.

Zavicefta is a combination of Avibactam sodium and Ceftazidime hydrate.

This study is seeking for patients with:

* sepsis (A very serious infection in your blood caused by germ (a bacteria)) or
* renal impairment (loss of kidney function) who are administrated with Zavicefta for the first time.

Subjects will take part in this study from the start date of receiving Zavicefta (Day 1) to Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received Zavicefta for the first time after the launch of Zavicefta
2. Patients who received Zavicefta for an infectious diseases indicated for Zavicefta
3. Patients with diagnosis of sepsis and/or renal impairment (creatinine clearance ≤ 50mL/min) at the start of the treatment with Zavicefta
4. Individuals who understand the nature of this study and give consent for the provision of the information collected in this study to third parties and the use of the information for other than intended use

Exclusion Criteria:

There are no exclusion criteria for this study.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with sepsis or renal impairment (creatinine clearance ≤ 50 mL/min) who are administrated with Zavicefta for the first time
Sampling Method: Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with adverse drug reactions (ADRs) | From the start date of the administration to 28 days after the administration (or 14 days after the date of discontinuation if the administration is discontinued)

SECONDARY OUTCOMES:
Number of Participants with Clinical Effectiveness | From the start date of the administration to 28 days after the administration (or 14 days after the date of discontinuation if the administration is discontinued)
Number of Participants with Clinical Effectiveness at the time of Test of Cure | 28 days after the start of the administration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3591038